CLINICAL TRIAL: NCT05334381
Title: Navigating Mental Health Treatment for Black Youth With Suicidal Risk
Brief Title: Navigating Mental Health Treatment for Black Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-019141; 1P50MH127511-01 (NIH)
Record Dates: First submitted 2022-04-05; First posted 2022-04-19 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Adolescent Behavior; Suicidal Ideation
Keywords: Youth Suicide; Cultural Adaptation; Mental Health Treatment; Health Disparities; Black Adolescents; Patient navigation
MeSH Terms: conditions — Adolescent Behavior; Suicidal Ideation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted STAT-ED (Experimental): The intervention will assist the family in following up with mental health referral recommendations provided by ED staff and eliciting families' preferences in regards to race and gender of providers, convenience of provider, and type of treatment. This assistance could involve help with the initial telephone contact, getting to appointments, and preparing for the appointments. The patient navigator will communicate with the family in person, by telephone, and/or by text messaging as per family's preference. This once to twice a week communication with both the youth and their parent will promote mental health care initiation and identify barriers and problem-solving solutions.
  Interventions: Behavioral: Adapted-STAT ED
- Standard Enhanced Treatment (Active Comparator): After discharge from the Children's Hospital of Philadelphia emergency department, the participant will be given a list of resources and referrals for mental health treatment by the hospital social work team. Phone call contact will be made to follow up on the initiation of treatment from the referral recommendations given at discharge.
  Interventions: Behavioral: Standard Enhanced Treatment

INTERVENTIONS:
Behavioral: Adapted-STAT ED — Patient navigator assigned to provide culturally informed motivational interviews, brief case management, psychoeducation and telephone contacts
  Arms: Adapted STAT-ED
Behavioral: Standard Enhanced Treatment — Follow up phone calls following discharge from the emergency department to confirm mental health treatment referral recommendations
  Arms: Standard Enhanced Treatment

SUMMARY:
This study looks to conduct a systematic adaptation of Suicidal Teens Accessing Treatment (STAT-ED) for Black youth presenting in the emergency department who have suicide risk. A randomized controlled trial of STAT-ED adapted for Black youth and their caregivers will examine whether patient navigation intervention can increase mental health treatment initiation and number of visits.

DETAILED DESCRIPTION:
Recent research has shown significant increases in suicides among Black youth and suicide attempts among Black high school students. Standard mental health treatment referrals were found to be not as effective among Black youth. This study in collaboration between Children's Hospital of Philadelphia and the University of Pennsylvania looks to determine if adapting standard Suicidal Teens Accessing Treatment (STAT-ED) to address barriers to initiating treatment for Black youth and their caregivers will increase mental health treatment initiation and number of treatment visits.

The primary objective is to conduct a systematic adaptation of STAT-ED for Black youth presenting in the emergency department who have suicidal risk. As well as to examine preliminary efficacy of the intervention on primary (mental health treatment initiation and number of visits) and secondary (suicidal ideation) outcomes using a prospective randomized controlled trial design.

The secondary objective is to examine implementation outcomes of adapted STAT-ED for Black youth and caregivers compared to enhanced treatment as usual.

Participants will be recruited from the Children's Hospital of Philadelphia emergency department and randomized to receive either adapted STAT-ED or enhanced treatment as usual following discharge from their emergency visit. 50 eligible youth and 50 eligible caregivers (50 youth-caregiver dyads) will be consented, enrolled, and randomized to produce 85 evaluable subjects. Treatment assignment will be done at the time of enrollment. Those chosen for the adapted STAT-ED will be assigned a patient navigator to provide culturally informed motivational interviews, assistance with appointments, barrier deduction discussions, and mental health information. The cultural adaptation will directly incorporate patients' preferences for treatment, such as treatment modalities, and address negative perceptions about treatment and stigma.

Descriptive statistics for demographics, motivation, suicidal ideation and affect will be measured at baseline. We will then assess use of treatment and services, motivation for treatment, suicidal ideation, and intervention acceptability at 2 months post-enrollment. At 6 months post-enrollment, the same measures as the 2 month follow-up will be assessed once more. The assessment scores will then be compared between the experimental and control treatment groups.

The results of this application would be expected to contribute important new knowledge on barriers faced by Black youth and their caregivers while initiating mental health treatment and examine if a culturally informed intervention will increase mental health treatment initiation.

ELIGIBILITY:
Youth Inclusion Criteria:

1. Identify as Black
2. Are between ages of 6-18 years
3. Endorse suicidal ideation and/or behaviors, or non-suicidal self harm within the last year at an ED or crisis response center visit
4. Live within Pennsylvania, Delaware, or New Jersey
5. Must be able to read and understand English

Youth Exclusion Criteria:

1. Does not identify Black as one of their races
2. Under 6 or over 18 years old
3. Does not speak English
4. No history of suicidal ideation, suicidal behavior, or non-suicidal self harm
5. Currently engaged in mental health treatment

Caregiver Inclusion Criteria:

1. Parent or legal guardian of eligible youth
2. Must be able to read and understand English

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Mental health treatment initiation | up to 6 months
  ED STARS mental health service use is a 8-item interview that measures mental health services children receive and actions taken by family to obtain services. This measure was used with over 6000 adolescents from the Pediatric Emergency Care Applied Research Network (PECARN) that spanned diverse geographic regions of the US (King et al., 2020). Cargeivers will complete this interview unless youth is participating without a parent.

SECONDARY OUTCOMES:
Suicidal ideation and behavior | up to 6 months
  Suicide Ideation Questionnaire-Junior (SIQ-Jr) is a youth report measure of frequency of suicidal thoughts over the last month.The SIQ-Jr is a 15-item questionnaire and is designed for students in Grades 7-9. Reliability coefficients are .93 to .94. SIQ-Jr has high internal consistency, test-retest reliability, predictive validity for suicidal behavior, and is sensitive to change.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda Boyd, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grupp-Phelan J, Stevens J, Boyd S, Cohen DM, Ammerman RT, Liddy-Hicks S, Heck K, Marcus SC, Stone L, Campo JV, Bridge JA. Effect of a Motivational Interviewing-Based Intervention on Initiation of Mental Health Treatment and Mental Health After an Emergency Department Visit Among Suicidal Adolescents: A Randomized Clinical Trial. JAMA Netw Open. 2019 Dec 2;2(12):e1917941. doi: 10.1001/jamanetworkopen.2019.17941. PMID 31860104
- [Background] King CA, Brent D, Grupp-Phelan J, Shenoi R, Page K, Mahabee-Gittens EM, Chernick LS, Melzer-Lange M, Rea M, McGuire TC, Littlefield A, Casper TC; Pediatric Emergency Care Applied Research Network (PECARN). Five Profiles of Adolescents at Elevated Risk for Suicide Attempts: Differences in Mental Health Service Use. J Am Acad Child Adolesc Psychiatry. 2020 Sep;59(9):1058-1068.e5. doi: 10.1016/j.jaac.2019.10.015. Epub 2019 Dec 9. PMID 31830523

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT05334381/Prot_SAP_001.pdf